CLINICAL TRIAL: NCT04766359
Title: Paclitaxel (Albumin-bound) Combined With Radiotherapy Compared With Cisplatin Combined With Radiotherapy for the Treatment of Early Stage Nasopharyngeal Carcinoma: a Prospective, Parallel-controlled, Multicenter Phase III Clinical Study
Brief Title: Paclitaxel (Albumin-bound) Combined With Radiotherapy for the Treatment of Early Stage Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yang Yang, Professor of medicine, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-236-02
Record Dates: First submitted 2021-02-14; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Albumin-Bound Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin-Bound paclitaxel combined with radiotherapy (Experimental): Albumin paclitaxel (100mg/m2), D1 intravenous drip, start the first week of radiotherapy, use it continuously for 4-6 weeks.
  Radiotherapy: The total dose is 66-70Gy, divided into 33-35 times to complete.
  Interventions: Drug: Albumin-Bound Paclitaxel
- Cisplatin combined with radiotherapy (Experimental): Cisplatin (40mg/m2), D1 intravenous drip, start the first week of radiotherapy, use it continuously for 4-6 weeks.
  Radiotherapy: The total dose is 66-70Gy, divided into 33-35 times to complete.
  Interventions: Drug: Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: Albumin-Bound Paclitaxel — Compare the effectiveness and safety of paclitaxel (albumin-bound) combined with radiotherapy and cisplatin combined with radiotherapy in the treatment of early nasopharyngeal carcinoma.
  Other Names: Cisplatin; Radiotherapy

SUMMARY:
This trial is a prospective, parallel controlled, randomized, open, multi-center phase III clinical trial. The trial will enroll 364 patients with nasopharyngeal carcinoma who are staged T1-2N0-1M0 (except T1N0M0) (UICC 8th edition) . This experiment was participated by multiple centers of Nanjing Gulou Hospital, Jiangsu Provincial People's Hospital, Jiangsu Cancer Hospital, Nanjing Military Region General Hospital, Jiangsu Provincial Hospital of Traditional Chinese Medicine, and Zhongda Hospital. Each center competes for admission of cases.

The subjects will be randomly assigned (using the random number table method according to the order of entry) to the experimental group to receive albumin-bound paclitaxel combined with IMRT concurrent radiotherapy, or the control group to receive cisplatin combined with IMRT concurrent radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Differentiated non-keratinizing carcinoma and undifferentiated non-keratinizing carcinoma confirmed by pathology;
* The staging is T1-2N0-1M0 (except T1N0M0) (UICC 8th edition);
* Initial treatment patients who have not received anti-tumor therapy;
* No history of other malignant tumors;
* Male or female, aged 18 to 70 years old;
* Liver and kidney function: total bilirubin ≤ upper limit of normal (ULN); AST and ALT ≤ 2.5 times ULN; alkaline phosphatase ≤ 5 times ULN; creatinine clearance ≥ 80 mL/min;
* Neutrophil count (ANC) ≥2×109/L, platelet count ≥100×109/L and hemoglobin ≥9 g/dL;
* No serious heart, lung, liver, kidney and other important organ dysfunction;
* Karnofsky score ≥70 points;
* Sign the informed consent form;
* Able to follow research protocols and follow-up procedures.

Exclusion Criteria:

* Anti-tumor treatment has been performed, including chemotherapy, radiotherapy, and surgery;
* Find distant metastases before treatment;
* Women who are pregnant or breastfeeding;
* Disagree to sign the informed consent form;
* Patients who cannot cooperate with regular follow-up due to psychological, social, family and geographic reasons;
* Simultaneously accept experimental treatment of other clinical research (in the treatment period of clinical research);
* Known to be allergic to possible chemotherapy drugs;
* Patients with other malignant tumors;
* Accompanied by severe uncontrollable infections or medical diseases, including autoimmune diseases;
* Major organ dysfunction, such as decompensated heart, lung, kidney, and liver failure, cannot tolerate radiotherapy and chemotherapy;
* Laboratory examination: total bilirubin>upper limit of normal (ULN); AST and/or ALT>1.5 times ULN and accompanied by alkaline phosphatase>2.5 times ULN;
* Any uncertain factors that affect patient safety or compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1month
  Nasopharyngeal + neck MRI and nasopharyngoscopy: the nasopharyngeal mass disappeared; the nasopharyngeal mucosa was smooth and no lesions were seen on the nasopharyngoscope. The tumor is clinically considered to have completely subsided. Neck MRI showed complete regression of cervical lymph nodes, or combined with clinical findings that the lymph node lesions completely resolved.